CLINICAL TRIAL: NCT06052891
Title: CHAMP For the Feeder: Pilot for CHAMP App Tube Weaning
Brief Title: CHAMP For the Feeder: Tube Feeding Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Lori Erickson (Other)
Collaborators: The Gerber Foundation (Other); Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor-Investigator, Lori Erickson, Director, Remote Health Solutions, Children's Mercy Hospital Kansas City
Organization: Children's Mercy Hospital Kansas City (Other)
Other Study IDs: STUDY00002775CMH
Record Dates: First submitted 2023-08-24; First posted 2023-09-25 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Feeding Disorders
Keywords: Pediatric; Feeding difficulties; Tube weaning
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: CHAMP Application — Children's Mercy Kansas City's CHAMP application was developed for data transfer of pediatric cardiac population vitals from home to the healthcare team in March 2014. CHAMP provides families and the clinical team with a new model of care leveraged by a remote patient monitoring (RPM) platform. CHAMP has been used in over 1000 patients, 28 states, and across 12 pediatric hospitals in pediatric cardiology. The CHAMP application is available in 11 languages for families to use on mobile devices (Apple and Android).

SUMMARY:
Single site evidence-based implementation of a mHealth application for remote patient monitoring for pediatric patients ready to wean from tube feedings (TFs). The primary objective of this study is to evaluate the CHAMP® ("CHAMP App") software platforms' expansion into TF weaning through Children's Mercy (CM) Kansas City's interdisciplinary feeding team (IDC). The investigators will use the current standard of care rates of tube weaning success, time to weaning, and healthcare team communication to evaluate the change after the implementation of the evidence-based CHAMP App. For equipoise of access, the study team will provide access in this pre-post design for parent/legally authorized representative (LAR)- child family access and use the CHAMP App software platform as soon as possible.

DETAILED DESCRIPTION:
Training: After consent to the study- parents/LAR will undergo training on the CHAMP App use by the study staff. The CHAMP App will be downloaded on the parent/LAR mobile device or an iPad that has been locked to contain only the CHAMP App and patient portal with mobile device management of the device by CM.

In addition to approval to begin a weaning trial by the IDC team providing primary nutrition management-beginning the weaning process may include these requirements:

* Weight for length or body mass index (BMI) must be stable. For children who are premature, syndromic, small for gestational age, or intrauterine growth restriction patients, this is at the dietitian's and provider's discretion. For typically developing patients, weight for length BMI z-score must be > -2.
* . Weekly feeding therapy is not required for tube weaning but will be strongly encouraged.
* A feeding therapist has assessed oral motor skills and agrees that the patient has sufficient skills to take all their calories by mouth.

CHAMP App use: Families will be provided with a weighing scale for home use; access to the CHAMP App mobile application or an iPad with the app and myChildren's Mercy App (patient portal) installed, if they prefer, during the study period. Data quality and validity will be ensured through the training of the healthcare team on data entry and out-of-range limits for each data value collected via the CHAMP web portal data entry forms. All data will be stored on the secure CM CHAMP Azure software platform with secure encryption database features.

Healthcare team CHAMP web portal use: The study team will review data entered by parents twice a week and as needed with questions and red flag concerns reported by parents/LAR. They will communicate back to parents with messages in the patient portal for documentation of messages that can be seen by other gastroenterology (GI) staff (GI clinic messages).

The IDC tube weaning algorithm (attached) will be used as a guideline for awareness of tube weaning but any changes to volume, concentration, or formula type will be reviewed and approved by an IDC provider before communicating to families.

RPM data entered by parents will be reviewed weekly by the IDC healthcare team in a team meeting organized through weekly reports of active patients enrolled in the study. This meeting will include an IDC provider, nurse, and nutritionist at minimum. There will be a summary of full study patient reports and individual patient reports available to all healthcare team members throughout the study, and these reports will be especially useful during these weekly meetings.

The IDC team works with Gastroenterology staff and fellows for 24 hours a day call. The CHAMP app will have a service pager for GI and the on-call hospital network is also available at any time for parents/LAR. On-call GI staff will be able to see feeding and weight data in Cerner under results review and CHAMP App. Videos are only available in the CHAMP web portal at champ.childrensmercy.org

Recommendation and timing for removal of feeding tubes will be up to the healthcare team alone. This event will be documented for date/time but is not a study-related intervention recommended through CHAMP App.

Additional measures to evaluate study results include:

Demographics - child and family measures: The study team will collect data on the child and family from the electronic medical record, including, but not limited to, infant medical conditions, feeding interventions, in-person healthcare visits with IDC and other specialists, language spoken, the distance of home residence from the hospital, in-home services used (Early Intervention, Physical Therapy, Occupational therapy, speech).

Nutritional measures: The study team will obtain the child's weight, length, and head circumference at birth and enrollment from the electronic medical record. The investigators will also obtain the following from the electronic medical record: weight for age and z-scores calculated by gender, weight percentiles, length/weight, mid-upper arm circumference (MUAC,) and head circumference. The investigators will use the CHAMP App to track weight at weekly intervals and obtain via parental report. There will be a weekly review, as well as on an as-needed basis, if sooner than weekly, by the IDC's research team, providers and nutrition team.

Healthcare team measures: The IDC team's periods of nutrition interventions will be evaluated for frequency of communication, including feeding interventions with families, volume changes, feeding routes, concentrations, and weight reporting frequency charted in the EMR. The time to first visit with the clinical team after referral to the IDC team, the rate of cancellation/no-show visits, and the number of patients on the wait list for enrollment in the clinical program will also be collected.

Family experience measures: Rate of first patient appointment attended, rate of attrition though never seen, cancellation and no-show appointments, time to first appointment after confirmation of visit in the calendar system, rate of follow-up frequency, graduation from the program with 100% calories by mouth with age-appropriate weight gain vs. attrition rates. Time to the healthcare recommendation of removal of feeding tube after the use of CHAMP app (by type nasogastric (NG) and gastrostomy - g-tube).

Technology measures by parents: Using the CHAMP App, the study team will track parent reported feeding volumes by mouth and tube, weights from home scales, videos of eating, and time to all feedings by mouth.

Technology adherence measures: The study team will track parent use of the app through tracking data on 1) app initiation, the first day of data transfer of CHAMP App data after enrollment; 2) implementation, the amount and type (feeding volumes, type, concentration, food amount, types, and weights) of asynchronous remote patient monitoring data received at the recommended intervals; and 3) discontinuation, the time of last data sent to the healthcare team.

ELIGIBILITY:
Eligibility Criteria: Parent/LAR-Child dyad was referred for feeding difficulty and tube feeding care at Children's Mercy.

* Inclusion Criteria

  * The child is between the ages of 1 month and five years 11 months.
  * Child is approved for a trial of tube weaning by the managing providers of their feeding difficulty.
* Exclusion Criteria

  * Children who do not meet the criteria to begin tube weaning.
  * Children who are older than 6 years of age at time of enrollment.
  * Parent/LAR of parent/LAR-child dyad who do not speak one of the languages offered via the CHAMP application (English, Spanish, German, Chinese, Vietnamese, Arabic, Korean, French, Filipino, Burmese or Somali).

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients in the Interdisciplinary Feeding Clinic (IDC) patient population that are deemed ready to begin weaning from tube feeds.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Adherence Initiation | Time in days, one event- the first day of data transfer of CHAMP App data after enrollment
  The study team will track parent use of the CHAMP App through tracking data on 1) app initiation the time of First data sent to the healthcare team.
Adherence Implementation | From enrollment to study endpoint, an average of 6 weeks
  The study team will track parent use of the CHAMP App through tracking data on implementation, the amount and type (feeding volumes, type, concentration, food amount, types (formula), and weights in kg) of asynchronous remote patient monitoring data received at the recommended intervals each week
Adherence Discontinuation | From enrollment to study endpoint, an average of 6 weeks
  The study team will track parent use of the CHAMP App through tracking data discontinuation at the time of last data sent to the healthcare team prior to completion of study activities.
Success rate to tube weaning | From enrollment to study endpoint, an average of 6 weeks
  Determine how the use of a remote patient monitoring mHealth software platform impacts the success rate (%) compared with those using only a standard outpatient interdisciplinary feeding tube using a tube weaning algorithm.
Time to weaning | From enrollment to study endpoint, an average of 4 weeks
  Determine how the use of a remote patient monitoring mHealth software platform the time (weeks) for children that were able to get 100% of calories by mouth while maintaining age-appropriate growth, compared with those using only a standard outpatient interdisciplinary feeding tube using a tube weaning algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Erickson, PhD, Principal Investigator — Children's Mercy Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Children's Mercy CHAMP Web Page — https://www.childrensmercy.org/about-us/remote-health-solutions/champ-app/